CLINICAL TRIAL: NCT01108237
Title: Comparison of In Vivo Alignment With TruMatch™ Personalized Solutions Compared to Conventional Instrumentation in Total Knee Replacement (TKR)
Brief Title: Alignment Comparison Between TruMatch™ Personalized Solutions and Conventional Total Knee Replacement Instrumentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08003
Record Dates: First submitted 2010-04-01; First posted 2010-04-21 (Estimated); Results first posted 2012-05-21 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Arthroplasties, Knee Replacement; Arthroplasties, Replacement, Knee; Arthroplasty, Knee Replacement; Knee Replacement Arthroplasties; Knee Replacement Arthroplasty; Knee Replacement, Total; Replacement Arthroplasties, Knee; Replacement Arthroplasty, Knee; Replacement, Total Knee; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TruMatch™ Personalized Solutions (Other): Cruciate Retaining and Posterior Stabilized Fixed-Bearing or Rotating Platform Total Knee Arthroplasty (PFC Sigma System) implanted using TruMatch™ Personalized Solutions
  Interventions: Other: TruMatch™ Personalized Solutions
- Historical Control (Other): Total Knee Arthroplasty (PFC Sigma System) implanted using conventional and CAS surgical techniques without TruMatch™ instrumentation.
  Interventions: Device: Total Knee Arthroplasty with Conventional Instrumentation.

INTERVENTIONS:
Other: TruMatch™ Personalized Solutions — TruMatch™ Personalized Solutions is the brand name of DePuy Orthopaedics, Inc. custom patient instrumentation. TruMatch™ is a pair of custom-made cutting blocks that allow distal femoral and proximal tibial cuts to be made according to a predefined surgical plan. The inner surface of the femoral block is manufactured to match the geometry of the patient's distal femur. The inner surface of the tibial block is manufactured to match the patient's proximal tibia. The geometric data is obtained from a CT scan and a preoperative plan approved by the surgeon.
  Arms: TruMatch™ Personalized Solutions
Device: Total Knee Arthroplasty with Conventional Instrumentation. — Total Knee Arthroplasty (PFC Sigma System) implanted using conventional instruments, not TruMatch™ instrumentation.
  Arms: Historical Control

SUMMARY:
This investigation is intended to provide clinical information about alignment using TruMatch™ and to compare the results to a conventional total knee replacement. TruMatch™ will be compared to a historical control study, which compares alignment results of computer aided surgery (CAS) and conventional surgical techniques.

The purpose of this investigation is to determine whether TruMatch™ alignment is non-inferior to alignment achieved with conventional instrumentation. This investigation will compare long leg alignment in total knee replacement achieved by the two types of procedures. Radiographic analysis will be performed by the same independent radiographic reviewer as the historical control study.

DETAILED DESCRIPTION:
The study is designed as a prospective, multi-center, non-randomized, clinical investigation to determine whether TruMatch™ alignment is non-inferior to alignment achieved in a recently completed study (historical control) with conventional instrumentation.

Each enrolled Subject will undergo a total knee replacement using the TruMatch™ surgical technique. This investigation will require the Subject to be followed once postoperatively to collect radiographs. Follow-up will occur typically 2 to 12 weeks after surgery and when the Subject can achieve full leg extension (+/-5 degrees) and can tolerate weight-bearing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following specific criteria will be considered for participation in the study:
* Subject is male or female and between the ages of 18 and 80 years old, inclusive.
* Subject requires a primary total knee replacement and is considered by the Investigator to be suitable for the specific knee prosthesis identified in the protocol.
* Subject has given voluntary, written informed consent to participate in this clinical investigation and has authorized the transfer of his/her information to DePuy.
* Subject has given consent to the transfer of his/her information to DePuy.
* Subject, who, in the opinion of the Clinical Investigator at the time of preoperative planning, are suitable for implantation using TruMatch™ instrumentation and whose surgical plan (patient proposal) is approved. For example, no femoral nails/bone plates that extend into the knee, i.e. within 8cm of joint line; no metal device that could cause CT scatter about the knee and no deformities greater than 15 degrees of fixed varus, valgus, or flexion

Exclusion Criteria:

* Subjects will be excluded from participation in the trial if they meet any of the following criteria:
* The Subject has, in the opinion of the Investigator, an existing condition that would compromise their participation and follow-up in this study.
* The Subject is a woman who is pregnant or lactating.
* The Subject is a known drug or alcohol abuser or has a psychological disorder that could affect follow-up care or treatment outcomes.
* The Subject has participated in a clinical investigation with an investigational product in the last 3 months.
* The Subject is currently involved in any personal injury litigation, medical-legal or worker's compensations claims.
* The Subject has previously had a prosthetic knee replacement device (any type including unicompartmental, total knee arthroplasty, patellofemoral arthroplasty) of the affected knee or a previous patellectomy.
* The Subject presents ankylosis of the hip joint on the side to be treated or previous ipsilateral UTO/HTO.
* The Subject requires simultaneous bilateral total knee replacements.
* The Subject had a contralateral TKA and that knee was previously entered in the study.
* Subject in whom the surgeon intends to implant a knee prosthesis that is not the cruciate retaining or posterior substituting PFC Sigma total knee arthroplasty.
* Subjects who have inflammatory arthritis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saleem Himden, BA, Study Director — DePuy Orthopaedics
Locations (4):
- United States (4):
  - Towson Orthopaedic Associates, Baltimore, Maryland
  - Summit Orthopaedics, LTD, Saint Paul, Minnesota
  - OrthoCarolina, Charlotte, North Carolina
  - Valley Orthopaedic Associates, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The TruMatch (patient-specific instruments) arm of this study was a prospective, multi-center, non-randomized, clinical investigation conducted at 4 sites. The other arm of this study (conventional instruments) included 86 historical control subjects.
Period: Overall Study
Arm/Group | TruMatch™ Personalized Solutions | Total Knee Arthroplasty With Conventional Instrumentation
Started | 73 (78 subjects were consented with intent to treat, however, 73 had surgery.) | 101
Completed | 64 (66 subjects underwent surgery per the protocol, however, only 64 met the primary end point.) | 86
Not Completed | 9 | 15
Not completed — No alignment data | 2 | 15
Not completed — Did not meet criteria for analysis | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TruMatch™ Personalized Solutions | Total Knee Arthroplasty With Conventional Instrumentation | Total
Number analyzed (Participants) | 66 | 86 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (8.4) | 64.6 (7.6) | 65.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 57 | 98
  Male | 25 | 29 | 54
Region of Enrollment [Count of Participants; unit: Participants]
  United States: United States | 66 | 86 | 152

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Axis Alignment(Absolute Value Measured in Degrees)Using 51 Inch Long Leg Films
Description: Limb alignment in TKR is important for accurate implant positioning. It is measured by looking at the mechanical axis of the limb. This axis is an imaginary line that starts at center of the femoral head and ends in the center of the talus. In a knee with normal alignment, this line (axis) passes near the joint center. Before surgery, the planned joint angle is recorded. This study measured the difference between the mechanical axis angle reached after surgery and the planned angle. Subjects with a mechanical alignment within 3 degrees of the planned angle were considered a success.
Time Frame: 12 weeks postoperatively (when subject has reached full knee extension)
Measure: Least Squares Mean (Standard Deviation); unit: Absolute value in degrees
Arm/Group | TruMatch™ Personalized Solutions | Total Knee Arthroplasty With Conventional Instrumentation
Number analyzed (Participants) | 64 | 84
Absolute value in degrees | 2.15 (1.85) | 2.14 (1.84)

2. Secondary Outcome: Compare Intraoperative Time Data During Procedure for Skin-to-skin Time in Minutes
Description: Intraoperative (skin to skin) time was measured to the nearest minute. TruMatch personalized Solutions and Conventional instrumentation outcomes are provided
Time Frame: During the Procedure
Population: Per protocol, to compare intraoperative time data, average skin to skin surgical time for knees, when using TruMatch and Conventional instrumentation
Measure: Mean (Standard Deviation); unit: Minutes
Units Other Than Participants: Knees
Groups:
- TruMatch Intraoperative Skin to Skin Time in Minutes: TruMatch intraoperative time in minutes during procedure
- Conventional Instrumentation Intraoperative Skin to Skin Time in Minutes: Intraoperative time during procedure in minutes for the skin to skin time
Arm/Group | TruMatch Intraoperative Skin to Skin Time in Minutes | Conventional Instrumentation Intraoperative Skin to Skin Time in Minutes
Number analyzed (Participants) | 66 | 86
Number analyzed (Knees) | 66 | 86
Minutes | 74.6 (15.3) | 79.8 (20.0)

3. Secondary Outcome: Tourniquet Time Measured in Minutes During the Procedure for TruMatch and Conventional Instruments
Description: Intraoperative Tourniquet time was measured to the nearest minute. TruMatch and Conventional instrumentation outcomes are provided
Time Frame: During the Procedure
Population: Per protocol, to compare intraoperative Tourniquet time data during knee replacement when using TruMatch and Conventional instrumentation
Measure: Mean (Standard Deviation); unit: Minutes
Units Other Than Participants: Knees
Groups:
- TruMatch Tourniquet Time in Minutes: TruMatch intraoperative Tourniquet time measured in minutes during knee procedure
- Conventional Instrumentation Tourniquet Time Measured in Minutes: Conventional Instrumentation Tourniquet time measured in minutes during knee procedure
Arm/Group | TruMatch Tourniquet Time in Minutes | Conventional Instrumentation Tourniquet Time Measured in Minutes
Number analyzed (Participants) | 66 | 86
Number analyzed (Knees) | 66 | 86
Minutes | 61.7 (16.3) | 60.5 (16.9)

4. Secondary Outcome: Tourniquet to 1st Bone Cut Measured in Minutes During the Procedure for TruMatch and Conventional Instruments
Description: Intraoperative Tourniquet to 1st Bone Cut time was measured to the nearest minute. TruMatch and Conventional instrumentation outcomes provided
Time Frame: During the Procedure
Population: Per protocol, to compare intraoperative Tourniquet time data during knee replacement when using TruMatch, Conventional instrumentation and Computer Assisted Surgery (CAS)
Measure: Mean (Standard Deviation); unit: Minutes
Units Other Than Participants: Knees
Groups:
- TruMatch Tourniquet to 1st Bone Cut Time in Minutes: TruMatch intraoperative Tourniquet to 1st Bone Cut time measured in minutes during knee procedure
- Conventional Instrumentation Tourniquet to 1st Bone Cut Time Measured in Minutes: Conventional Instrumentation Tourniquet to 1st Bone Cut time measured in minutes during knee procedure
Arm/Group | TruMatch Tourniquet to 1st Bone Cut Time in Minutes | Conventional Instrumentation Tourniquet to 1st Bone Cut Time Measured in Minutes
Number analyzed (Participants) | 64 | 85
Number analyzed (Knees) | 64 | 85
Minutes | 9.0 (2.5) | 10.3 (4.0)

5. Secondary Outcome: Coronal Alignment Femoral and Tibial
Description: Femoral Component to mechanical axis (degrees) and Tibial component to mechanical axis (degrees)
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Femoral Component to Mechanical Axis / TruMatch: Femoral component to mechanical axis (degrees) TruMatch at 3-months
- Femoral Component to Mechanical Axis Conventional: Femoral component to mechanical axis (degrees) Conventional at 3-months
- Tibial Component to Mechanical Axis TruMatch: Tibial component to mechanical axis (degrees) for TruMatch at 3-months
- Tibial Component to Mechanical Axis Conventional: Tibial component to mechanical axis (degrees) for Conventional at 3-months
Arm/Group | Femoral Component to Mechanical Axis / TruMatch | Femoral Component to Mechanical Axis Conventional | Tibial Component to Mechanical Axis TruMatch | Tibial Component to Mechanical Axis Conventional
Number analyzed (Participants) | 66 | 86 | 66 | 86
Degrees | 89.8 (1.3) | 90.0 (1.7) | 90.0 (1.1) | 90.5 (1.9)

6. Secondary Outcome: Sagittal Component Alignment
Description: Sagittal Component Alignment analyzed and reported at 3- months
Time Frame: Collected at Pre-Op, 3 months
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Femoral Sagittal Component Alignment TruMatch: Femoral Sagittal Component Alignment for TruMatch Cohort at 3-months (Femoral Component Flexion in degrees)
- Femoral Sagittal Alignment Conventional: Femoral Sagittal Alignment Conventional TKA at 3-months (Femoral Component Flexion in degrees)
- Tibial Sagittal Alignment TruMatch: Sagittal Alignment TruMatch / Tibial Posterior Slope (degrees) at 3-months
- Tibal Sagittal Alignment Conventional: Sagittal Alignment Conventional / Tibial Posterior Slope (degrees) at 3-months
Arm/Group | Femoral Sagittal Component Alignment TruMatch | Femoral Sagittal Alignment Conventional | Tibial Sagittal Alignment TruMatch | Tibal Sagittal Alignment Conventional
Number analyzed (Participants) | 64 | 86 | 64 | 86
Degrees | 90.1 (2.5) | 89.8 (2.2) | 88.5 (2.8) | 86.7 (2.7)

ADVERSE EVENTS:
Arm/Group | TruMatch™ Personalized Solutions | Total Knee Arthroplasty With Conventional Instrumentation
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/84
Other Adverse Events (participants affected / at risk) | 0/64 | 17/84
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TruMatch™ Personalized Solutions (N=64) | Total Knee Arthroplasty With Conventional Instrumentation (N=84)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 17 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less